CLINICAL TRIAL: NCT04081779
Title: IMPACT: Improving Access to Cancer Survivorship Via Telehealth
Brief Title: Survivorship Care Plans and Telehealth Education for the Improvement of Access to Cancer Survivorship, the IMPACT Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RG1005815; NCI-2019-05726 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10267 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); R21CA258105 (NIH)
Record Dates: First submitted 2019-08-29; First posted 2019-09-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Breast Carcinoma; Colorectal Carcinoma; Lung Carcinoma; Lymphoma; Prostate Carcinoma
Keywords: Cancer survivors; survivorship care plans; primary care
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Lymphoma; Prostatic Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods; Palliative Care

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: Personnel other than the statisticians and lay health educators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Arm I (patient-generated SCP) (Active Comparator): Patients receive a self-generated SCP (i.e., generated from baseline questionnaire responses).
  Interventions: Other: Survivorship Care Plan; Other: Questionnaire Administration
- Arm II (patient-generated SCP, counseling) (Experimental): Patients receive a self-generated SCP as in Arm I. Patients also receive a 30-minute telephone-based educational counseling session on survivorship care administered by trained lay health counselors.
  Interventions: Other: Survivorship Care Plan; Other: Educational Intervention; Other: Questionnaire Administration
- Arm III (generic information) (Active Comparator): Patients receive generic information on survivorship care on study.
  Interventions: Other: Questionnaire Administration; Other: Supportive Care
- Arm IV (generic information, patient-generated SCP) (Active Comparator): Patients receive generic information on survivorship care and a self-generated SCP as in Arm I on study.
  Interventions: Other: Survivorship Care Plan; Other: Questionnaire Administration; Other: Supportive Care
- Arm V (generic information, patient-generated SCP, counseling) (Experimental): Patients receive generic information on survivorship care as well as a self-generated SCP as in Arm I and a telephone-based educational counseling session as in Arm II on study.
  Interventions: Other: Survivorship Care Plan; Other: Educational Intervention; Other: Questionnaire Administration; Other: Supportive Care

INTERVENTIONS:
Other: Survivorship Care Plan — Receive patient-generated SCP
  Arms: Arm I (patient-generated SCP); Arm II (patient-generated SCP, counseling); Arm IV (generic information, patient-generated SCP); Arm V (generic information, patient-generated SCP, counseling)
Other: Educational Intervention — Receive telephone-based educational counseling session
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm II (patient-generated SCP, counseling); Arm V (generic information, patient-generated SCP, counseling)
Other: Questionnaire Administration — Ancillary studies
Other: Supportive Care — Receive generic information on survivorship care
  Other Names: Supportive Therapy; Symptom Management
  Arms: Arm III (generic information); Arm IV (generic information, patient-generated SCP); Arm V (generic information, patient-generated SCP, counseling)

SUMMARY:
This trial studies how well self-generated survivorship care plans and telehealth education works in improving knowledge and self-efficacy in cancer survivors living in rural areas. Patients living in rural areas often face barriers to survivorship care and report unmet needs. A survivorship care plan created by the patient (self-generated) may help them to better transition from oncology to primary care and improve communication between care teams in order to meet these needs and create better health outcomes. Telehealth is a way of delivering health care services from a distance, including patient education. Combining a self-generated survivorship care plan with telehealth education may help to improve knowledge and self-efficacy in cancer survivors.

DETAILED DESCRIPTION:
OUTLINE:

Patients complete a questionnaire at baseline (paper, online, or telephone-based) and have medical records reviewed and are assigned to 1 of 3 cohorts.

COHORTS A AND B: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive a self-generated SCP (i.e., generated from baseline questionnaire responses).

ARM II: Patients receive a self-generated SCP as in Arm I. Patients also receive a 30-minute telephone-based educational counseling session on survivorship care administered by trained lay health counselors.

COHORT C: Patients are randomized to 1 of 3 arms.

ARM III: Patients receive generic information on survivorship care on study.

ARM IV: Patients receive generic information on survivorship care and a self-generated SCP as in Arm I on study.

ARM V: Patients receive generic information on survivorship care as well as a self-generated SCP as in Arm I and a telephone-based educational counseling session as in Arm II on study.

PRIMARY CARE PROVIDERS: Primary care providers complete a questionnaire about perceptions of the SCP and self-efficacy in providing survivorship care.

ONCOLOGY CLINICS: Participants complete Organizational Readiness to Change Assessment (ORCA) questionnaire and participate in a qualitative interview about perceptions of implementation of survivorship care.

After completion of study, patients are followed up at approximately 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Cancer survivors who have completed curative therapy within the past 5 years (may still currently be on long-term/targeted non-cytotoxic agent maintenance therapy, e.g., tamoxifen or aromatase inhibitors for breast cancer survivors; androgen deprivation therapy for prostate cancer survivors)
* History of either adult-onset (age >= 18) lymphoma, breast, colorectal, lung, or prostate cancer
* Able to perform all study requirements, including responding to questionnaires
* Willing to be randomized
* Capable of providing informed consent
* Consent to release oncology and primary care medical records
* English or Spanish speakers
* PRIMARY CARE PROVIDERS: PCPs responsible for delivering primary care to IMPACT study participants will be contacted about participating in the study after participant enrollment into the study.
* ONCOLOGY STAFF: Oncology Staff (Oncologists, Nurse Practitioners, Physician's assistants) will be recruited from sites involved in the IMPACT study
* CLINIC ADMINISTRATORS: Clinic administrators will be recruited from sites involved in the IMPACT study

Exclusion Criteria:

* Currently on palliative or hospice care, or considering transferring to such care within the next 3 months
* Lacks telephone access
* Lacks mailing address or ability to receive study materials electronically
* Currently being followed in a pediatric clinical setting (either for primary care or for cancer care)
* History of having had > 1 cancer type diagnosed and treated (exception is for skin cancers treated with surgical excision alone; also, individuals who only have had relapse of their initial cancer remain eligible so long as they have completed curative therapy and meet all other eligibility criteria)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Initial participation rate of cancer survivors identified from community-based or partner practices, and Cancer Surveillance System of Western Washington | Up to 8 weeks
Accuracy of survivors' self-generated survivorship care plans (SCPs) in relation to those based on medical record abstraction | Up to 8 weeks
  Will measure the accuracy of participants' SCPs by comparing their self-reported medical history collected via questionnaire, with data abstracted from medical records. Accuracy will be reported by percentage of missing data in the self-generated SCP compared to medical records, and percentage of incorrect data in the self-generated SCP compared to medical records.
Proportion of survivors who receive the phone-based education session within the study time period | Up to 8 weeks
Proportion of survivors who complete the follow-up questionnaire within the study time period | Up to 8 weeks
Response rate among primary care providers (PCPs) to the PCP survey | Up to 8 weeks

SECONDARY OUTCOMES:
Participant perceived self-efficacy: questionnaire using the PROMIS Global 10 and health related self-efficacy scales | Up to 8 weeks
  The effects of the intervention versus (vs.) control on participant perceived self-efficacy will be measured at baseline and at the end of the study via a questionnaire using the PROMIS Global 10 and health related self-efficacy scales.
Survivorship knowledge | Up to 8 weeks
  The effects of the intervention vs. control on survivorship knowledge will be measured at baseline and at the end of the study via a questionnaire.
PCP self-efficacy towards survivorship care | Up to 8 weeks
  The effects of the intervention vs. control on PCP self-efficacy towards survivorship care will be measured at baseline and at the end of the study via a questionnaire using the PROMIS Global 10 and health related self-efficacy scales.
Local oncology clinics' attitudes towards survivorship care implementation | Up to 8 weeks
  Assess oncology practitioners' and clinic administrators' views on utility and feasibility of implementing SCPs in target clinics, using the ORCA (Organizational Readiness to Change Assessment) instrument and qualitative interviewing

CONTACTS AND LOCATIONS:
Overall Officials: Eric Chow, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yi JC, Lee E, Duggan C, Baker KS, Blythe N, Cole AM, Cushing-Haugen KL, Gutierrez AI, Linden H, Mendoza JA, Ohlsen TJD, Ortblad KF, Schwartz SM, Yung R, Ceballos R, Chow EJ. Perspective of Hispanic Cancer Survivors on Survivorship Care Plans: A Qualitative Study. J Immigr Minor Health. 2025 Oct 14. doi: 10.1007/s10903-025-01794-8. Online ahead of print. PMID 41087806
- [Derived] Chow EJ, Blythe NA, Cushing-Haugen KL, Duggan C, Baker KS, Cole AM, Green S, Guiterrez AI, Lee E, Linden HM, Mendoza JA, Ohlsen TJD, Ortblad KF, Schwartz SM, Yung RL, Ceballos RM. Enhancing survivorship care among Hispanic/Latino cancer survivors via lay health educators: results of a pilot randomized trial. J Cancer Surviv. 2025 Feb 15:10.1007/s11764-025-01758-9. doi: 10.1007/s11764-025-01758-9. Online ahead of print. PMID 39955465
- [Derived] Duggan C, Cushing-Haugen KL, Cole AM, Allen J, Gilles R, Hornecker JR, Gutierrez AI, Warner J, Baker KS, Ceballos RM, Chow EJ. Feasibility of delivering survivorship care via lay health educators: A pilot randomized controlled trial among rural cancer survivors. J Rural Health. 2023 Jun;39(3):666-675. doi: 10.1111/jrh.12736. Epub 2023 Jan 2. PMID 36593127

DOCUMENTS (1):
  • Informed Consent Form (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT04081779/ICF_001.pdf